CLINICAL TRIAL: NCT04949126
Title: Self Medication and Pulpal and Periapical Dental Pain
Brief Title: Self Medication in Odontology (AUDE)
Acronym: AUDE
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2021 COUSSON; 2021-A00417-34 (Other: ANSM)
Record Dates: First submitted 2021-06-18; First posted 2021-07-02 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2023-06

CONDITIONS: Dental Anxiety; Dental Pain
Keywords: Anxiety; Pulpal pain; Self medication; Observational study
MeSH Terms: conditions — Toothache; Anxiety Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- acute pain of pulpal origin: no intervention
  Interventions: Behavioral: questionnaire
- anxious group: no intervention
  Interventions: Behavioral: questionnaire

INTERVENTIONS:
Behavioral: questionnaire — questionnaires of precarity, dental anxiety, self medication, pain

SUMMARY:
To describe and understand the self-medication behaviours of a population of adults coming to the Clermont-Ferrand dentistry department for acute pain of pulpal origin and of a population of adults coming to the specific care unit of the Clermont-Ferrand dentistry department or the Riom hospital for treatment under general anaesthesia.

DETAILED DESCRIPTION:
Self-medication behaviour will be studied by means of a questionnaire. Questionnaires on insecurity, anxiety about dental care, items related to the ingestion function of the International Classification of Functioning, Disability and Health (ICF), a visual analogue pain assessment scale and the PCS-CF pain dramatisation scale will also be used.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient, male or female, coming to consult in the Clermont-Ferrand or Riom Hospital for acute pain of pulp origin and periapical OR eligible for dental treatment under general anesthesia in a context phobic.
* Understanding and practicing French
* giving informed consent to participate in research.
* Affiliation to a Social Security scheme.

Exclusion Criteria:

* Patients under guardianship.
* Patient's refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient with acute pain of pulp origin and periapical or eligible for dental treatment under general anesthesia in a context phobic.
Sampling Method: Non-Probability Sample
Enrollment: 940 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
description of the self-medication behaviours | day 0
  evaluated by patient interrogation

SECONDARY OUTCOMES:
level of anxiety | day 0
  : evaluated with IDAF 4C (anxiety module between 8-40, phobia module between 5-10 and anxious situations between 10 and 50), the higher the score, the more anxious the patient is
level of insecurity | day 0
  evaluated by questionnaire (EPICES (the patient is in situation of insecurity if the score is higher than 30))
description of the oral health with the related to the ingestion function of the International Classification of Functioning, Disability and Health (ICF) | day 0
  each item is evaluated with a Lickert scale
visual analogue pain assessment scale and the PCS-CF pain dramatisation scale | Day 0
  PCS-CF scale is evaluated between 0 and 52, the higher the score, the more patient is over reacting faced with pain

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Yves Cousson, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France